CLINICAL TRIAL: NCT03891459
Title: Neural Account of Social Placebo Effect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Normal University (Other)
Responsible Party: Principal Investigator, ma, yina, Principal Investigator, Beijing Normal University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: FSPE
Record Dates: First submitted 2019-03-17; First posted 2019-03-27 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Spray+ Group; Control Group
Keywords: social placebo effect; fMRI; neural account
MeSH Terms: interventions — Behavior Control

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- spray+ group (Experimental): In spray+ condition, participants learned oxytocin materials on a self-paced basis and then intranasally administered with saline (but it was told as "oxytocin"). Participants were instructed to refrain from smoking or drinking (except water) for 2 h before the experiment. The spray was administered to each participant three times, and each administration consisted of one inhalation into each nostril. Participants took a rest (they were told it was a time period waiting for treatment to produce effects) for 10min and then performed the experimental tasks.
  Interventions: Behavioral: spray+ manipulation
- control group (Placebo Comparator): In control condition, the materials and procedure were same with the spray+ condition except the nasal spray was told as "saline" instead. Oxytocin materials used in current experiments were adopted from previous study
  Interventions: Behavioral: control manipulation

INTERVENTIONS:
Behavioral: spray+ manipulation — Participants in spray+ group received placebo manipulation and were told they sprayed was oxytocin (in fact, it was saline);
  Arms: spray+ group
Behavioral: control manipulation — Participants in control group were told they sprayed saline (in fact, it was saline).
  Arms: control group

SUMMARY:
The current study aimed to reveal the neural mechanism of social placebo belief formation and belief representation, and also investigated how the brain pattern predict the social behavior performance under placebo manipulation.

DETAILED DESCRIPTION:
Participants were randomly assigned to spray+ group (sprayed with saline but told as "oxytocin") and control group (sprayed with saline but told as "saline"). After 10 min, participants were invited to the resting-state, text viewing task in fMRI scanner.

In resting state session, participants with their eyes open and were instructed to attend to a black fixation cross centrally presented on a grey projection screen for 8 min (240TR).

The Text viewing task employed a mixed block and even-related fMRI design. Participants were asked to judge whether they could understand the stimuli or not by a button press (1=understand; 2=not understand). Three kinds of stimuli were presented in separate block including "oxytocin-function", "oxytocin-knowledge", "robot" related stimuli, each category contained 20 sentences. In each block, the sentence (within one category) was presented pseudo-randomized from 5s to 9s (with mean duration of 7s), then followed by a jittered time interval (interval time = sentence duration - response time; if participants made response within 5s, the sentence would not disappear until its duration reached 5s). There were two sessions with six blocks per session, and there were 5 sentences (trials) per block. The order of blocks and sentences were designed to present in pseudo-random order and were applied to all participants.

ELIGIBILITY:
Inclusion Criteria:

* All participants had normal or corrected-to-normal vision, and mental healthy.

Exclusion Criteria:

* Participants who reported no history of neurological, endocrine or psychiatric disorders, who majored in psychology in college or recently participated in any other drug study were not recruited.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 68 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2018-11-05 (Actual)

PRIMARY OUTCOMES:
The brain functional connectivity | 8 mins, 240 TR in scanner
  For functional connectivity estimation, we adopted DLPFC, mPFC and reward related brain regions as the seeds to do whole-brain connectivity analysis. And the conducted two-sample T test to examine whether there would be some differences between spray+ and control groups.
Social brain network properties in resting-state | 8 mins, 240 TR in scanner
  For the network properties, we chose the social brain network as our target and interested network, then estimated the global efficiency within this network.And the conducted two-sample T test to examine whether there would be some differences between spray+ and control groups.
The brain response pattern for the key concepts about oxytocin | 5.33mins, 160TR in scanner
  We estimated the beta response trial by trial for each single concept and then investigated the neural representation of all concepts by using representational similarity analysis (RSA).

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Normal University, Beijing, Beijing Municipality, China